CLINICAL TRIAL: NCT04279353
Title: Effectiveness of Mindfulness Based Intervention (MBI) Technique in Reducing Stress Levels of Anesthesiology and Intensive Therapy Residents at the Faculty of Medicine, University of Indonesia
Brief Title: Effectiveness of Mindfulness Based Intervention in Reducing Stress Levels of Anesthesiology and Intensive Therapy Residents at the Faculty of Medicine, University of Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Amir S Madjid, Professor, MD, PhD, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IndonesiaUAnes 045
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Anesthesiology and Intensive Therapy Residents at the Faculty of Medicine, University of Indonesia
Keywords: Stress, Resident, Anesthesiologist, Mindfulness, Medical, Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Based Intervention (Experimental): Participants was asked to answer PSS-10 questionnaire to measure their stress level, then they received Mindfulness Based Intervention program for 4 weeks and did the PSS-10 test again after 4 weeks.
  Interventions: Other: Mindfulness Based Intervention

INTERVENTIONS:
Other: Mindfulness Based Intervention — this intervention is a 4 weeks program with logbook and follow up during intervention

SUMMARY:
This study was conducted to determine the effectiveness of MBI technique in reducing the stress level of anesthesiology and intensive therapy residents at the Faculty of Medicine, University of Indonesia.

DETAILED DESCRIPTION:
This research was an experimental study with paired one group design. The research subjects were anesthesiology and intensive therapy residents at the Faculty of Medicine, University of Indonesia in 2019. The MBI program lasted four weeks, consisted of one formal face-to-face training and informal training through homework carried out every day for four weeks. 13 study subjects met the inclusion criteria and did not enter the exclusion criteria. 1 study subject must be excluded because it did not complete the informal training. Data collection on the Perceived Stress Scale 10 Item (PSS-10) was conducted in July and August 2019.

ELIGIBILITY:
The inclusion criteria for participation were being anesthesiology and intensive therapy resident stationed in Cipto Mangunkusumo Hospital, having a PSS-10 score ≥ 14, and agreeing to fully participate in the study.

The exclusion criteria for this study were: (1) residents who used narcotic/psychotropic drugs during the study period and (2) residents who were not able to complete the study or attend the formal face-to-face training as scheduled due to conflicting work schedule.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
PSS-10 test | 30 minutes test
  this is a test to measure stress level

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gurman GM, Klein M, Weksler N. Professional stress in anesthesiology: a review. J Clin Monit Comput. 2012 Aug;26(4):329-35. doi: 10.1007/s10877-011-9328-7. Epub 2011 Dec 17. PMID 22180163
- [Result] Alexander BH, Checkoway H, Nagahama SI, Domino KB. Cause-specific mortality risks of anesthesiologists. Anesthesiology. 2000 Oct;93(4):922-30. doi: 10.1097/00000542-200010000-00008. PMID 11020740
- [Result] De Hert S. Burnout Among Anesthesiologists: It׳s Time for Action! J Cardiothorac Vasc Anesth. 2018 Dec;32(6):2467-2468. doi: 10.1053/j.jvca.2018.06.010. Epub 2018 Jun 19. No abstract available. PMID 30093191
- [Result] Hutchinson TA, Haase S, French S, McFarlane TA. Stress, Burnout and Coping among Emergency Physicians at a Major Hospital in Kingston, Jamaica. West Indian Med J. 2014 Jun;63(3):262-6. doi: 10.7727/wimj.2013.330. Epub 2014 Jun 12. PMID 25314285
- [Result] West CP, Dyrbye LN, Erwin PJ, Shanafelt TD. Interventions to prevent and reduce physician burnout: a systematic review and meta-analysis. Lancet. 2016 Nov 5;388(10057):2272-2281. doi: 10.1016/S0140-6736(16)31279-X. Epub 2016 Sep 28. PMID 27692469